CLINICAL TRIAL: NCT01125527
Title: A Phase III Observer-blind, Randomized, Controlled, Single-coordinating Center Study to Investigate Immunogenicity and Safety of a Monovalent Glycoprotein-conjugated (Diptheria Toxin -CRM197) Hib Vaccine in 13-59 Months Old Healthy Children in China, According to the Recommended Regimen of 1 Dose
Brief Title: Immunogenicity and Safety of a Monovalent Glycoprotein-Conjugated (Diptheria Toxin -CRM197) Hib Vaccine in 13-59 Months Old Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V37_06
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2011-12

CONDITIONS: Haemophilus Influenzae Type b (Hib) Infection
Keywords: Haemophilus influenzae type b (Hib); Vaccine; Anti PRP antibody
MeSH Terms: conditions — Haemophilus Infections; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Biological: Monovalent glyco-conjugated vaccine against Haemophilus influenzae type b (Hib)
- Arm 2 (Active Comparator)
  Interventions: Biological: Tetanus toxoid polysaccharide-conjugated vaccine against Haemophilus influenzae type b (Hib)

INTERVENTIONS:
Biological: Monovalent glyco-conjugated vaccine against Haemophilus influenzae type b (Hib) — a single dose was administered
  Arms: Arm 1
Biological: Tetanus toxoid polysaccharide-conjugated vaccine against Haemophilus influenzae type b (Hib) — a single dose was administered
  Arms: Arm 2

SUMMARY:
This study will evaluate the safety and immunogenicity of single dose of two commercially available vaccines used to prevent Haemophilus influenzae type b infections in children 13-59 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants 13-59 months of age.

Exclusion Criteria:

* Prior Hib vaccine administration.
* History of serious reaction(s) following vaccination.
* Any vaccination within 7 days of study vaccination.
* Known or suspected immune impairment.
* Premature (before 37th week of gestation) or birth weight less than 2500g
* For additional entry criteria please refer to the protocol.

Ages: 13 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Anti-PRP antibody levels at day 31 post last vaccination | 30 days after last vaccination

SECONDARY OUTCOMES:
Solicited local and systemic reactions, AEs, and SAEs | 30 days post last vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Province, China